CLINICAL TRIAL: NCT00400868
Title: A Randomized Controlled Study to Evaluate the Short- and Long-term Effectiveness of an Individualized Resource Oriented Occupational Therapy for Patients With Rheumatoid Arthritis
Brief Title: Effectiveness of Occupational Therapy in Patients With Rheumatoid Arthritis(RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Zürcher Rheumastifung, Zurich, Switzerland (Other); Gertrude and Wolfgang Schrader Dislich Foundation (Other); Swiss Ligue Against Rheumatism, Zurich, Switzerland (Unknown)
Responsible Party: Karin Niedermann, MPH, University Hospital Zurich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: niedk_EK444_
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis, occupational therapy, joint protection
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (1):
- standard joint protection education (Active Comparator): psycho-educational joint protection vs. usual care (standard joint protection education)
  Interventions: Behavioral: psycho-educational Joint protection education

INTERVENTIONS:
Behavioral: psycho-educational Joint protection education — individualized psycho-educational joint protection education, 4-times over 3 weeks; one additional booster session 2 months later

SUMMARY:
The purpose of the study is to compare the short- and long-term effectiveness of an individualized, resource-oriented joint protection intervention with the standard, problem-oriented joint protection intervention for patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Joint Protection (JP)is an important intervention in the management of people with arthritis. Altering working methods (e.g. use of proximal joints, dynamic activities), energy conservation (balance between activity and rest) and using assistive devices should place less strain on joint structures weakened by the disease process. These strategies ought to decrease pain and stress on joints, improve function, and facilitate maintaining social roles.

The effectiveness of JP has been evaluated in a number of studies, all in a group setting. JP has beneficial short-term effects on pain and function in patients with established RA and moderate functional problems. Using assistive devices reduces pain during task performance in comparison to normal methods and altering working methods significantly reduces difficulties in activities of daily living (ADL). However this generally does not result in significant behavioral changes and a long-term impact on reducing pain and maintaining function may only be reached if JP is taught using behavioral education methods. Additionally, adherence of RA patients to different interventions is generally modest, which may well determine the effectiveness of any given intervention, especially in the long-term.

All previous studies were carried out in group settings, however, in Switzerland, standard JP education is provided on a one-to-one basis and an individualized education is assumed to be a promising approach.

This clinical trial aims to test the hypothesis that an individualized, resource-oriented JP education in RA patients leads to a better therapy success in the short and long-term, compared to problem-oriented standard JP education in terms of joint protection behavior. Secondary outcome parameters are self-perception, general and specific self-efficacy and general and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to ACR Guidelines (1988)
* Actual hand pain on activity or history of wrist and/or metacarpophalangeal(MCP) joint pain and inflammation
* Referred to OT for a Joint Protection intervention program
* Willingness to comply with the randomly assigned treatment and informed consent
* Functional Class: 2 to 4
* German speaking/understanding/reading
* Sufficient cognitive capacities to understand the aims and procedures of the proposed study and the requirements of participation

Exclusion Criteria:

* Functional class 1 (anticipated self-exclusion, as patients in class 1 will not be referred to JP).
* Severe finger, hand, elbow or shoulder deformities
* Insufficient ability to understand, speak and read the German language
* Insufficient cognitive capacities to understand the aims and procedures of the proposed study and the requirements of participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
joint protection behavior | before/after intervention, 3,6,12 months follow up

SECONDARY OUTCOMES:
General quality of life | before intervention, 3,6,12 months follow up
Health related quality of life / physical functional ability | before intervention, 6,12 months follow up
Self-Illness Separation SIS, derived from the PRISM (intervention group) | before/during/after intervention, 3,6,12 months follow up
Goals achievement (intervention group) | during/after intervention, 3,6,12 months follow up
Hand impairment status, including pain | before/during/after intervention, 3,6,12 months follow up
Arthritis self-efficacy and JP-specific self-efficacy | before/after intervention, 3,6,12 months follow up
Self-perceived disease activity | before intervention, 12 months follow up
Clinical data | before intervention, 3, 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Robert de Bie, Prof, PhD, Study Director — University of Maastricht NL; Karin Niedermann, MPH, Principal Investigator — University Hospital of Zurich, CH; Stefan Buchi, MD, Study Director — University Hospital of Zurich, CH
Locations (4):
- Switzerland (4):
  - University Hospital, Bern
  - Rehabilitation Clinic, Valens
  - Schulthess Klinik, Zurich
  - University Hospital, Zurich